CLINICAL TRIAL: NCT00958971
Title: A Multi-center, Open Label Phase II Trial of TKI258 in FGFR1 Amplified and Non-amplified Metastatic or Advanced HER2 Negative Breast Cancer
Brief Title: Safety and Efficacy of TKI258 in FGFR1 Amplified and Non-amplified Metastatic HER2 Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2202; 2008-006430-10 (EudraCT Number)
Record Dates: First submitted 2009-08-11; First posted 2009-08-14 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-09

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast cancer; HER2 negative; FGFR1
MeSH Terms: conditions — Breast Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TKI258 - Positive (Experimental): These are the participants who had a positive T(4;14) status
  Interventions: Drug: TKI258
- TKI258 - Negative (Experimental): These are the participants who had a negative T(4;14) status
  Interventions: Drug: TKI258
- TKI258 Non-interpretable (Experimental): These are the participants who had a non-interpretable T(4;14) status
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258 — All participants received a singly daily oral dose of 500 mg dovitinib on a 5 days on/2 days off schedule in 28 cycles.
  Other Names: Dovitinib

SUMMARY:
The purpose of this trial is to determine the efficacy and safety profile of TKI258 in 3 groups of patients with metastatic HER2 negative breast cancer (BC) stratified by FGFR1 and hormone receptor (HR) status.

ELIGIBILITY:
Inclusion Criteria:

1. Female presenting with metastatic breast cancer.
2. Tumor must have been tested by FISH/CISH for FGFR1 amplification.
3. HER2 and HR status must have been determined.
4. Patients must have HER2 negative breast cancer.
5. Patients must have a documented disease progression as define by RECIST at baseline.
6. Patients with HR+ disease:

   * Must have received at least one prior endocrine therapy in the metastatic setting.
   * Must have received no more than three lines of chemotherapy in the metastatic setting.
7. Patients with HR- disease must have received at least one and no more than three lines of chemotherapy in metastatic setting.

Exclusion Criteria:

1. Patients with known brain metastases or who have signs/symptoms attributable to brain metastases and have not been assessed with radiologic imaging to rule out the presence of brain metastases.
2. Impaired cardiac function or clinically significant cardiac diseases, including any of the following:

   * History or presence of serious uncontrolled ventricular arrhythmias or presence of atrial fibrillation.
   * Clinically significant resting bradycardia (< 50 beats per minute).
   * LVEF assessed by 2-D echocardiogram (ECHO) or Multiple gated acquisition scanning (MUGA)< 45%.
3. Any of the following within 6 months prior to study entry: myocardial infarction (MI), severe/unstable angina, Coronary Artery Bypass Graft (CABG), Congestive Heart Failure (CHF), Cerebrovascular Accident (CVA), Transient Ischemic Attack (TIA), Pulmonary Embolism (PE).
4. Uncontrolled hypertension defined by a SBP > 150mm Hg and/or DBP > 100mm Hg, with or without anti-hypertensive medication.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-07; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Complete responses (CR) or partial response (PR) defined according to RECIST | Every 8 weeks

SECONDARY OUTCOMES:
Clinical Benefit (CR, PR and SD ≥ 24 weeks after start of study treatment), PFS | Every 8 weeks
Safety and tolerability of TKI258 treatment assessed by frequency and severity of Adverse Events. | Monthly
Pharmacokinetic: plasma concentrations and PK parameters (e.g. Cmax, Tmax, AUC0-t) | Study Day 1, 5 , 26, 52, 78

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (37):
- United States (18):
  - Comprehensive Blood and Cancer Center Dept CBCC (3), Bakersfield, California
  - Tower Cancer Research, Beverly Hills, California
  - UCLA/ University of California Los Angeles Div. of Hematology/Oncology, Los Angeles, California
  - Cancer Care Associates Medical Group Dept. of CCA, Redondo Beach, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Florida Cancer Specialists Dept.of FloridaCancerSpec. (2), Fort Myers, Florida
  - Kansas City Cancer Center KCCC (3), Overland Park, Kansas
  - Associates in Oncology/Hematology, P.C., Rockville, Maryland
  - Comprehensive Cancer Centers of Nevada, Henderson, Nevada
  - UNC/ Lineberger Comprehensive Cancer Center Dept. of Linberger Cancer Ctr, Chapel Hill, North Carolina
  - Northwest Cancer Specialists Northwest Office (2), Portland, Oregon
  - Texas Oncology, P.A. Dept. of Texas Oncology, Bedford, Texas
  - Texas Oncology, P.A. Austin, Dallas, Texas
  - Texas Oncology, P.A. Presbyterian Hospital, Dallas, Texas
  - Texas Oncology, P.A. Texas Oncology - Sammons, Dallas, Texas
  - Tyler Cancer Center Dept.ofTylerCancerCtr. (2), Tyler, Texas
  - Fairfax Northern Virginia Hematology Oncology Fairfax NVH, Fairfax, Virginia
  - Blue Ridge Research Center at Roanoke Neurological Center Blue Ridge Cancer Care, Roanoke, Virginia
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Montreal, Quebec
- Novartis Investigative Site, Helsinki, Finland
- France (4):
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Saint-Herblain Cédex
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Villejuif
- Italy (6):
  - Novartis Investigative Site, Cuneo, CN
  - Novartis Investigative Site, Cremona, CR
  - Novartis Investigative Site, Parma, PR
  - Novartis Investigative Site, Candiolo, TO
  - Novartis Investigative Site, Napoli
  - Novartis Investigative Site, Negrar
- Spain (3):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Lleida, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Taipei, Taiwan
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, London

REFERENCES:
- See also: Results for CTKI258A2202 from the Novartis Clinical Trials website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=5425